CLINICAL TRIAL: NCT02239913
Title: Topiramate-Phentermine Combinations for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Professor, University of Kentucky
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED IN 27; R01DA032254 (NIH)
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine; Pharmacotherapy; Phentermine; Topiramate; Self-Administration
MeSH Terms: interventions — Cocaine; Phentermine; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Subjects will be maintained on placebo and phentermine during placebo maintenance. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo; Drug: Phentermine
- Topiramate Dose 1 (Experimental): Subjects will be maintained on the low topiramate dose. Subjects will be maintained on placebo and phentermine during maintenance on the low dose of topiramate. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo; Drug: Phentermine; Drug: Topiramate
- Topiramate Dose 2 (Experimental): Subjects will be maintained on the high topiramate dose. Subjects will be maintained on placebo and phentermine during maintenance on the high dose of topiramate. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo; Drug: Phentermine; Drug: Topiramate

INTERVENTIONS:
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and topiramate.
Drug: Placebo — The pharmacodynamic effects of placebo will be determined during maintenance on placebo and topiramate.
Drug: Phentermine — The pharmacodynamic effects of phentermine maintenance will be determined during maintenance on placebo and topiramate.
  Other Names: Adipex®
Drug: Topiramate — The pharmacodynamic effects of chronic topiramate will be determined.
  Other Names: Topamax®
  Arms: Topiramate Dose 1; Topiramate Dose 2

SUMMARY:
This study will determine the influence of topiramate (Topamax®) and phentermine (Adipex®), alone and in combination, on the reinforcing, subjective and physiological effects of cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use by the intranasal or intravenous route

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine, topiramate or phentermine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Reinforcing Effects | Nine times over approximately five weeks inpatient admission.
  The reinforcing effects of cocaine will be determined using a self-administration procedure in which subjects choose to take previously sampled doses.

SECONDARY OUTCOMES:
Subjective effects | Nine times over approximately five weeks inpatient admission.
  Subjects will complete subjective effects measures during nine sessions while they are admitted to our inpatient unit. These items will ask about drug effects and general mood.
Physiological Effects | Daily over approximately five week inpatient admissions
  Physiological measures will be completed daily while subjects are admitted to our inpatient unit. Physiological measures include temperature, heart rate and blood pressure.
Side effects | Daily over approximately five weeks of inpatient admission
  Subjects will complete a side effects questionnaire daily while they reside on the inpatient unit. Side Effects questions will query subjects about common effects of centrally active medications.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Rush, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States